CLINICAL TRIAL: NCT01764399
Title: Care4U: Self Management Intervention for Older Adult Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0552-12-FB
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Risk Factor
Keywords: cardiovascular risk factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care4U intervention (Experimental): Care4U intervention with 6 weekly sessions focusing on physical activity, healthy eating, self-management, emotional responses.
  Interventions: Behavioral: Care4U
- Information group (No Intervention): The information group receives 6 weekly socialization sessions.

INTERVENTIONS:
Behavioral: Care4U
  Arms: Care4U intervention

SUMMARY:
Older adults caring for others often neglect their own health. This research is being done to see if helping caregivers focus on their own needs can improve their health and ability to care for others

DETAILED DESCRIPTION:
The specific aims are to evaluate the Care4U intervention in order to refine the intervention for a larger clinical trial, which includes 1) subject acceptability of the intervention, 2) evaluation of intervention delivery, fidelity, and data collection, and 3) evaluation of the components of the intervention (patient activation, knowledge, self-efficacy, and CV self-management strategies).

Recruitment was conducted in 2 acute care hospitals from April 2013 through Dec 2013. Six caregivers were enrolled during this time, with one dropping out after baseline.

The participants completing the study (n=5) provided data related to the aim. Four participants were able to use Adobe Connect via the provided laptops with written instructions and phone coaching. Delivery of the intervention via Adobe connect was enjoyed by the participants, with minimal connectivity problems. Participants were interested in websites and videos related to their health, but did not relate exploring these links on the laptop desktop without suggestion from the PI.

ELIGIBILITY:
Inclusion Criteria:

* Describes self as an informal Caregiver of patient who has undergone cardiac surgery (revascularization, valve, or combination)and performs ≥1 activity of daily living or instrumental activity of daily living for the patient
* ≥ 65 years
* Self-reports ≥1 modifiable cardiovascular risk (hypertension, hyperlipidemia, physical inactivity, obesity)
* Lives in the same residence with patient
* Oriented to person, place, and time (asking the subject to state their name, where he/she is (for example what building, town and state) and what time it is (time, day, date)
* Able to hear, and speak and read English

Exclusion Criteria:

* Permanent residence in skilled or assisted care facility
* Participation in 3 times per week exercise during the past 6 months. -

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity | Baseline, 6 weeks, and 3 months
  Physical activity will be measured via self-report and with Actigraphy.

SECONDARY OUTCOMES:
Change in healthy diet intake | Baseline, 6 weeks, 3 months
  Change in self-reported diet intake
Change in emotional functioning (stress, anxiety, depression) | Baseline, 6 weeks, 3 months
  Change in self-reported stress, anxiety and depression scores

CONTACTS AND LOCATIONS:
Overall Officials: Paula S Schulz, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Bryan Health, Lincoln, Nebraska, United States